CLINICAL TRIAL: NCT03317457
Title: A Randomized Phase II Study of Durvalumab (MEDI4736) and Tremelimumab Compared to Doxorubicin in Patients With Advanced or Metastatic Soft Tissue Sarcoma
Brief Title: Durvalumab and Tremelimumab Compared to Doxorubicin in Patients With Advanced or Metastatic Soft Tissue Sarcoma
Acronym: MEDISARC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AIO-Studien-gGmbH (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AIO-STS-0415; 2016-004750-15 (EudraCT Number)
Record Dates: First submitted 2017-10-18; First posted 2017-10-23 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Metastatic Adult Soft Tissue Sarcoma; Recurrent Adult Soft Tissue Sarcoma
MeSH Terms: conditions — Sarcoma | interventions — durvalumab; tremelimumab; Doxorubicin

STUDY DESIGN:
Intervention Model Description: Treatment Arm A: Combination of Durvalumab and Tremelimumab Treatment Arm B: Doxorubicin
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Durvalumab and Tremelimumab (Experimental): Cycles/courses 1-3:
  Durvalumab 1.5g q4wks Tremelimumab 75 mg q4wks
  Cycles/courses ≥4:
  Durvalumab 1.5g q4wks Tremelimumab 75 mg q12wks
  Interventions: Biological: Durvalumab and Tremelimumab
- Doxorubicin (Active Comparator): Doxorubicin 75 mg/qm q3wks for 6 courses
  Interventions: Drug: Doxorubicin

INTERVENTIONS:
Biological: Durvalumab and Tremelimumab — immun checkpoint inhibitor
  Arms: Durvalumab and Tremelimumab
Drug: Doxorubicin — Anthracycline
  Arms: Doxorubicin

SUMMARY:
The objective of the trial is to assess the efficacy of Durvalumab and Tremelimumab in comparison to doxorubicin in treatment-naïve Soft tissue sarcoma patients

ELIGIBILITY:
Inclusion Criteria:

* 1. Written informed consent and any locally-required authorization (EU Data Privacy Directive in the EU) obtained from the subject prior to performing any protocol-related procedures, including screening evaluations 2. Age ≥ 18 years at time of study entry 3. Body weight > 30kg at study inclusion 4. Histologically confirmed diagnosis of metastatic or advanced soft tissue sarcoma of intermediate or high grade [according to FNCLCC score; intermediate=grade 2 score of 4-5 points, high grade = grade 3 score of 6-8 points] with disease progression within 6 months prior to study inclusion:

  • Fibrosarcoma

  • Pleomorphic high grade sarcoma ("malignant fibrous histiocytoma")

  • Leiomyosarcoma
  * Liposarcoma (myxoid liposarcoma, dedifferentiated liposarcoma, pleomorphic liposarcoma)
  * Malignant glomus tumor
  * Rhabdomyosarcoma, alveolar or pleomorphic (excluding embryonal)
  * Vascular sarcoma (angiosarcoma)
  * Synovial sarcoma
  * High-grade sarcoma, not otherwise specified (NOS)
  * Malignant peripheral nerve sheath tumors
  * Other types of sarcoma (not listed as ineligible), if approved by the coordinating investigator / study coordinator.

Excluding:

Uncertain differentiation (epithelioid, alveolar soft part, clear cell, desmoplastic small round cell, malignant mesenchymoma, PEComa), chondrosarcoma, Ewing sarcomas/PNET, chordoma, malignant solitary fibrous tumors, embryonal rhabdomyosarcoma, osteosarcoma, gastrointestinal stromal tumors, dermatofibrosarcoma protuberans, inflammatory myofibroblastic sarcoma (low-grade), neuroblastoma, malignant mesothelioma, and mixed mesodermal tumors of the uterus (Study inclusion is based on local histopathological diagnosis). 5. Metastatic or locally advanced STS, not amendable to surgery with curative intention.

6. No prior treatment line for advanced or metastatic disease. 7. ECOG performance status 0-2 8. Patients with measurable disease (at least one uni-dimensionally measurable target lesion by CT-scan or MRI) according to Response Evaluation Criteria in Solid Tumors (RECIST 1.1) are eligible.

9. If prior palliative radiotherapy has been given to metastatic lesions: either ≥1 measurable lesion remains outside the radition field or the sole lesion meets RECIST 1.1 criteria for progression at study entry.

10. Patients with bone lesions as the only measurable lesion are eligible, provided that lesions consist of soft tissue, which is measurable via CT or MRI.

11. Prior radiotherapy and surgery are allowed if completed 4 weeks (for minor surgery and palliative radiotherapy for bone pain: 2 weeks) prior to start of treatment and patient recovered from toxic effects.

12. Adequate blood count, liver-enzymes, and renal function:

* Haemoglobin ≥ 9.0 g/dL
* Absolute neutrophil count (ANC) ≥ 1.5 x 109/L (> 1500 per mm3)
* Platelet count ≥ 100 x 109/L (>100,000 per mm3)
* Serum bilirubin ≤ 1.5 x ULN. This will not apply to subjects with confirmed Gilbert's syndrome (persistent or recurrent hyperbilirubinemia that is predominantly unconjugated in the absence of hemolysis or hepatic pathology), who will be allowed only in consultation with their physician.
* AST (SGOT)/ALT (SGPT) ≤ 2.5 x institutional upper limit of normal unless liver metastases are present, in which case it must be ≤ 5x ULN
* Serum creatinine CL>40 mL/min by the Cockcroft-Gault formula (Cockcroft and Gault 1976) or by 24-hour urine collection for determination of creatinine clearance 13. Adequate cardiac function (left ventricular ejection fraction ≥50% as assessed by ECHO) 14. Female subjects must either be of non-reproductive potential (ie, post-menopausal by history: ≥60 years old and no menses for ≥1 year without an alternative medical cause; OR history of hysterectomy, OR history of bilateral tubal ligation, OR history of bilateral oophorectomy) or must have a negative serum pregnancy test upon study entry.

  15. Subject is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up.

Exclusion Criteria:

* 1. Patients who are suitable for anthracycline-based combination therapies 2. Cardiac events such as arrhythmias, myocardial infarction, CHF, apoplexy, lung embolism within 6 months prior to study treatment 3. Mean QT interval corrected for heart rate (QTc) ≥470 ms calculated from 3 electrocardiograms (ECGs) using Fredericia's correction 4. Uncontrolled severe hypertension (failure of diastolic blood pressure to fall below 100 mmHg and systolic blood pressure >160 mmHg) 5. Previous malignancy (other than STS) which either progresses or requires active treatment.

Exceptions are: basal cell cancer of the skin, pre-invasive cancer of the cervix, T1a or T1b prostate carcinoma, or superficial bladder tumor [Ta, Tis and T1].

6. History or clinical evidence of CNS metastases

Exceptions are: Subjects who have completed local therapy and who meet both of the following criteria:

1. are asymptomatic and
2. have no requirement for steroids 6 weeks prior to start of study treament. Screening with CNS imaging (CT or MRI) is required only if clinically indicated or if the subject has a history of CNS metastases 7. Active or prior documented autoimmune disease within the past 2 years. NOTE: Subjects with vitiligo, Grave's disease, or psoriasis not requiring systemic treatment (within the past 2 years) are not excluded.

   8. Active or prior documented inflammatory bowel disease (e.g., Crohn's disease, ulcerative colitis) 9. History of primary immunodeficiency 10. History of allogeneic organ transplant 11. History of hypersensitivity to durvalumab, tremelimumab (alone or in combination), doxorubicin or any of the constituents of the products 12. Medication that is known to interfere with any of the agents applied in the trial.

   13. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, active peptic ulcer disease or gastritis, active bleeding diatheses including any subject known to have evidence of acute or chronic hepatitis B, hepatitis C or human immunodeficiency virus (HIV), or psychiatric illness/social situations that would limit compliance with study requirements or compromise the ability of the subject to give written informed consent.

   14. Major surgical procedure (as defined by the Investigator) within 28 days prior to the first dose of study medication. Note: Local surgery of isolated lesions for palliative intent is acceptable.

   15. Any unresolved toxicity >CTCAE grade 2 from previous anti-cancer therapy with the exception of alopecia, vitiligo, and the laboratory values defined in the inclusion criteria.
   * Patients with Grade ≥2 neuropathy will be evaluated on a case-by-case basis after consultation with the Coordinating Investigator.
   * Patients with irreversible toxicity not reasonably expected to be exacerbated by treatment with durvalumab or tremelimumab (if applicable) may be included only after consultation with the Coordinating Investigator.

     16. Any prior Grade ≥3 immune-related adverse event (irAE) while receiving any previous immunotherapy agent, or any unresolved irAE >Grade 1 17. Known history of previous clinical diagnosis of tuberculosis 18. Receipt of live attenuated vaccination within 30 days prior to study entry or within 30 days of receiving durvalumab 19. Female subjects who are pregnant, breast-feeding or male or female patients of reproductive potential who are not employing an effective method of birth control (failure rate of less than 1% per year) 20. Any condition that, in the opinion of the investigator, would interfere with evaluation of study treatment or interpretation of patient safety or study results 21. Participation in another clinical study with an investigational product during the last 30 days before inclusion 22. Any previous treatment with a PD-1 or PD-L1 or CTLA-4 inhibitor, including durvalumab and tremelimunab 23. Current or prior use of immunosuppressive medication within 28 days before the first dose of durvalumab, with the exceptions of intranasal and inhaled corticosteroids or systemic corticosteroids at physiological doses, which are not to exceed 10 mg/day of prednisone, or an equivalent corticosteroid 24. Receipt of the last dose of anti-cancer therapy (chemotherapy, immunotherapy, endocrine therapy, targeted therapy, biologic therapy, tumor embolization, monoclonal antibodies, other investigational agent) ≤ 21 days prior to the first dose of study drug or ≤4 half-lifes of the agent administered, which ever comes first.

     25. Previous enrollment or randomization in the present study (does not include screening failure).

     26. Patient who has been incarcerated or involuntarily institutionalized by court order or by the authorities (§ 40 Abs. 1 S. 3 Nr. 4 AMG).

     27. Patients who are unable to consent because they do not understand the nature, significance and implications of the clinical trial and therefore cannot form a rational intention in the light of the facts [§ 40 Abs. 1 S. 3 Nr. 3a AMG].

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2017-12-15 (Actual); Primary Completion 2022-08-12 (Actual); Study Completion 2022-08-12 (Actual)

PRIMARY OUTCOMES:
overall survival (OS) | up to 57 months from randomization

SECONDARY OUTCOMES:
AEs / SAEs and Treatment Emergent Adverse Events according to CTCAE 4.03 | up to 18 months from randomization
  Assessment of adverse events of tremelimumab and durvalumab (MEDI4736) combination therapy
Objective Response Rate (ORR) according to RECIST 1.1 criteria | up to 57months from randomization
OS mile stone rate at 24 months | up to 24 months from randomization
Duration of response | up to 57 months from randomization
progression-free survival (PFS) | up to 57 months from randomization
Quality of life QLQ-C30 | up to 12 months from randomization
  scores according to EORTC QLQ-C30 scoring manual (Quality of life)

CONTACTS AND LOCATIONS:
Overall Officials: Viktor Grünwald, Dr., Principal Investigator — Universitätsklinikum Essen
Locations (1):
- Medizinische Hochschule Hannover, Hanover, Germany

IPD SHARING:
Plan to Share IPD: No